CLINICAL TRIAL: NCT04978753
Title: Phase II Clinical Study of the Efficacy and Safety of Anlotinib Combined With Almonertinib in the First-line Treatment of Patients With Brain Metastases From EGFR Mutation-positive Non-small Cell Lung cancer-----a Prospective, Single-arm Exploratory Study
Brief Title: the Efficacy and Safety of Anlotinib Combined With Almonertinib in the First-line Treatment of Patients With Brain Metastases From EGFR Mutation-positive Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li-kun Chen (Other)
Responsible Party: Sponsor-Investigator, Li-kun Chen, sun yat-sen university cancer center, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO 1063
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Non-small Cell Lung Cancer; Brain Metastases
Keywords: EGFR mutation; NSCLC; brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — anlotinib; aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): Anlotinib (12mg/time (BSA≥1.6 m2) or 10mg/time (BSA<1.6 m2), once a day orally, taking two weeks and stopping for one week) combine with Almonertinib (110mg, orally once a day)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — 1. Anlotinib: 12mg/time (BSA≥1.6 m2) or 10mg/time (BSA<1.6 m2), once a day orally, taking two weeks and stopping for one week;
  2. Almonertinib: 110mg, orally once a day;
  Other Names: almonertinib

SUMMARY:
Subject population：Patients with brain metastases from EGFR mutation-positive non-small cell lung cancer who have not received systemic treatment.

Experimental design: Single-center, single-arm phase II clinical trial. Purpose: Efficacy and safety of Anlotinib combined with Almonertinib in the treatment of patients with brain metastases from EGFR mutation-positive non-small cell lung cancer.

treatment plan: 1). Anlotinib: 12mg/time (BSA≥1.6 m2) or 10mg/time (BSA<1.6 m2), once a day orally, taking two weeks and stopping for one week; 2). Almonertinib: 110mg, orally once a day; primary endpoint: Intracranial progression-free survival (iPFS); secondary endpoint: Objective intracranial response rate (iORR=iCR+iPR), intracranial disease control rate (iDCR=iCR+iPR+i SD), overall progression-free survival (PFS), overall survival (OS), quality of life score.

ELIGIBILITY:
Inclusion Criteria:

1) 18-75 years old, ECOG PS score: 0-2 points; and there is no worsening of the disease within 2 weeks before enrollment, and the expected survival time is more than 3 months; 2) Advanced non-small cell lung cancer diagnosed by histology or cytology; 3) Baseline inspection confirms that the tumor has EGFR sensitive mutations (first-generation or second-generation sequencing, the detection can accept the following two types of tissue: archive tumor tissue; tumor tissue freshly collected during the screening period); 4) Asymptomatic or mildly symptomatic brain metastases (headache, nausea or epilepsy and other symptoms can be controlled with a fixed dose of mannitol/dexamethasone/pain relievers/antiepileptic drugs for more than 3 days); 5) MRI confirmed tumor metastasis to brain parenchyma, brain lesions ≥3; or patients with 1-2 brain lesions but not suitable for local treatment or refusal to local treatment. The brain lesions must have at least one measurable lesion with a diameter of ≥5mm; 6) Have not received systemic treatment after brain metastasis (the treatment adopted by neoadjuvant treatment is not included in the treatment plan, and the recurrence within 6 months after the end of the adjuvant treatment, the adjuvant treatment part is defined as first-line treatment, and cannot be included in this study; If the recurrence is more than 6 months, adjuvant treatment will not be included in the treatment plan); 7) The main organs are functioning normally, that is, they meet the following standards:

1. The standard of routine blood examination must meet (no blood transfusion within 14 days, no use of granulocyte colony stimulating factor and other hematopoietic stimulating factors):
2. HB≥90g/L;
3. ANC≥1.5×109/L;
4. PLT ≥80×109/L;
5. The biochemical inspection shall meet the following standards:
6. TBIL <1.5 times the upper limit of normal (ULN);
7. ALT and AST<2.5 ULN; if there is liver metastasis, ALT and AST<5 ULN;
8. Cr≤1.25 ULN or creatinine clearance (CCr) ≥45ml/min (Cockcroft-Gaulat formula);
9. Urine protein <2+ (when the baseline urine protein is 2+, a 24-hour urine protein quantification should be performed, and it can only be selected when it is ≤1g);
10. The international normalized ratio of blood coagulation (INR) ≤ 1.5 and APTT ≤ 1.5 ULN;
11. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%); 8) Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; serum or urine pregnancy test is negative within 7 days before study entry , And must be non-lactating patients; men should agree to patients who must use contraception during the study period and within 6 months after the end of the study period.

9) The patients voluntarily joined the study, signed an informed consent form, and had good compliance.

Exclusion Criteria:

1) Small cell lung cancer (including lung cancer mixed with small cell carcinoma and non-small cell carcinoma); 2) Brain metastases accompanied by active bleeding; 3) Those who have previously used anti-tumor angiogenesis drugs (such as bevacizumab, endurance, anlotinib, etc.) treatment failure; 4) At the beginning of the study treatment, there was an unhealed toxic reaction of grade ≥2 (NCI-CTC AE4.03) related to the previous treatment: (except for hair loss and grade 2 neuropathy caused by platinum drugs) 5) Those who have a variety of factors that affect oral medications (such as uncontrollable nausea and vomiting, inability to swallow, gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.); 6) Local radiotherapy to relieve the disease within 14 days before the first administration of the study treatment; radiotherapy or extensive radiotherapy for more than 30% of the bone marrow area within 4 weeks before the first administration (for palliative treatment of non-brain metastases such as bone metastases) Except for radiotherapy); 7) Patients with any severe and/uncontrolled diseases, including:

1. Patients with unsatisfactory blood pressure control (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
2. Meet any of the following cardiac standards: In the resting state, the average corrected QT interval (QTcF) obtained from 3 ECG examinations is ≥470 msec (Fredericia formula is used, see Appendix 4 for details). Various clinically significant heart rhythm, conduction, and resting ECG morphological abnormalities, such as complete left bundle branch block, third-degree block, second-degree block, and PR interval ≥250 msec. Various factors that may increase the risk of QTc prolongation or the risk of arrhythmia events, such as cardiac insufficiency according to NYHA standards III to IV; heart failure; hypokalemia; congenital long QT syndrome; family history with long first-degree relatives QT syndrome or sudden death of unknown cause under 40 years of age; various combined medications that may prolong the QT interval.
3. Active or uncontrolled serious infection;
4. Liver diseases such as cirrhosis, decompensated liver disease, chronic active hepatitis;
5. Poor diabetes control (fasting blood glucose (FBG)> 10mmol/L);
6. Urine routine shows that urine protein is ≥++, and the 24-hour urine protein quantification is confirmed to be greater than 1.0 g; 8) Long-term unhealed wounds or fractures; 9) Pulmonary hemorrhage with NCI CTC AE grade> Grade 1 occurred within 4 weeks before enrollment; other parts of bleeding with NCI CTC AE grade> Grade 2 occurred within 4 weeks before enrollment; hemorrhage tendency (such as active peptic ulcer) Or patients who are receiving thrombolytic or anticoagulant therapy such as warfarin, heparin or their analogues; 10) Those who have had arterial/venous thrombotic events within 12 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; 11) Clinically significant hemoptysis (more than 50ml of hemoptysis per day) occurred within 3 months before enrollment; or significant clinically significant bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood at baseline ++ and above, or suffer from vasculitis, etc.; 12) Have the following past history: interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy, clinically active interstitial lung disease; 13) People who have a history of psychotropic drug abuse and cannot be quit or have mental disorders; 14) Respiratory syndrome (≥CTC AE grade 2 dyspnea), severe pleural fluid, ascites, and pericardial effusion; 15) A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; active infection, such as HBV (HBV DNA copy number> 103/ml), HCV, HIV, etc.; 16) According to the judgment of the investigator, those with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.

17) The patient has active ingredients or inactive excipients, chemical structure and AZD9291 (and/or anlotinib) to AZD9291 (and/or anlotinib) A history of hypersensitivity to drugs similar to / or Anlotinib or AZD9291 (and/or Anlotinib).

18) Men or women who have fertility but have not taken effective contraceptive measures, women are pregnant or breastfeeding, or have a positive pregnancy test (urine or serum) before entering the study.

19) Because the patient is unwilling to comply with the research procedures, restrictions and requirements, the researcher determines that the patient should not participate in the research.

20) Allogeneic bone marrow transplantation has been performed. 21) Any serious or uncontrolled eye disease may increase the safety risk of the patient according to the judgment of the investigator; 22) In the 120 days before the collection of genetic samples, whole blood without leukocytes was transfused; 23) The patient has other coexisting malignant tumors or has been diagnosed with other malignant tumors in the last 5 years, except for basal cell carcinoma, cervical or squamous cell skin cancer in situ, and papillary thyroid carcinoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
iPFS | 10-25months
  Intracranial progression-free survival

SECONDARY OUTCOMES:
iORR | 10-25momths
  Objective intracranial response rate
iDCR | 10-25months
  intracranial disease control rate
PFS | 10-25momths
  overall progression-free survival
OS | 10-40months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Likun Chen, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Pan Y, Li M, Yu H, Zhang B, Yu M, Hou X, Chen L. Efficacy and safety with aumolertinib plus anlotinib for untreated EGFR-mutant NSCLC with brain metastases. NPJ Precis Oncol. 2025 Dec 1;10(1):2. doi: 10.1038/s41698-025-01191-2. PMID 41326640